CLINICAL TRIAL: NCT05474872
Title: Postoperative Delirium: a Complex Prediction Model in Patients Undergoing Major Abdominal Surgery
Brief Title: Postoperative Delirium in the ICU Setting of an Eastern European Centre
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Responsible Party: Principal Investigator, Mara Sonia Mihaescu, Principal Investigator, PhD Student, Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor
Other Study IDs: 456/12.01.2022
Record Dates: First submitted 2022-07-23; First posted 2022-07-26 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Delirium; Cognitive Impairment
Keywords: postoperative delirium; abdominal surgery; malondialdehyde; S100B protein; Tau protein; pNF-H; Bispectral Index; anesthesia depth; general anesthesia
MeSH Terms: conditions — Emergence Delirium; Cognitive Dysfunction; Frontotemporal Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood collected for serum analysis of biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BIS monitoring: Patients in this group will be subjected to Bispectral index-guided general anesthesia.
  Interventions: Device: BIS monitoring
- PRST score monitoring: Patients in this group will be subjected PRST score-guided general anesthesia.

INTERVENTIONS:
Device: BIS monitoring — The depth of anesthesia will be monitored using Bispectral Index values.
  Groups: BIS monitoring

SUMMARY:
The study targets postoperative delirium in patients undergoing major abdominal surgery, with the aim to evaluate the functional baseline and proteomics implicated in pathogenesis, prevention strategies (such as anesthesia depth monitoring) and incidence in certain population groups.

ELIGIBILITY:
Inclusion Criteria:

* ASA risk I-III;
* patients undergoing complex digestive surgery, such as esophagectomy, total gastrectomy, hemicolectomy, cephalic duodenopancreatectomy, hepatic resection.

Exclusion Criteria:

* the impossibility of obtaining the patient's consent/his decisional incapacity;
* patients who underwent neurosurgery for cerebrospinal lesions / cardiac surgery under cardiopulmonary bypass;
* prediagnosed senile/vascular/mixed dementia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 to 70 years, given informed consent, who will be subjected to major abdominal surgery and admitted in the ICU postoperatively, will be assessed from the preoperative period until hospital discharge, to collect the requisite information.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Prediction model for postoperative delirium (POD) in major abdominal surgery | 3-4 years
  Developing an accesible algorithm to anticipate the occurence of postoperative delirium, based on functional baseline and proteomics, in adult patients subjected to major abdominal surgical interventions.
  This includes investigating a correlation between a set of risk factors, a panel of biomarkers and the occurrence of postoperative delirium in the enrolled patients, respectively.

SECONDARY OUTCOMES:
Anesthesia depth monitoring and the incidence of postoperative delirium | 0-4 days postoperatively
  Assessing the influence of BIS monitoring during general anesthesia on the prevalence of postoperative delirium
Postoperative delirium incidence in surgical patients in the Intensive Care Unit (ICU) setting | during ICU hospitalization
Postoperative delirium incidence in surgical patients - subgroup - communism survivors | during ICU hospitalization
Postoperative delirium incidence in surgical patients - subgroup - patients with no relatives/visitors | during ICU hospitalization

OTHER OUTCOMES:
The influence of POD on length of stay (LOS), unplanned ICU re-admission, cognitive decline and mortality | during patient hospitalization
  Evaluating the possibility of a correlation between the occurence of POD and prolonged hospitalization, a prerequisite for ICU re-admittance or further cognitive deterioration / mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ionescu, MD, PhD, Study Director — Regional Institute of Gastroenterology and Hepatology Prof. Dr. O. Fodor; Mara Mihaescu, PhD student, Principal Investigator — Regional Institute of Gastroenterology and Hepatology Prof. Dr. O. Fodor
Locations (1):
- Regional Institute of Gastroenterology and Hepatology "Prof.Dr.O.Fodor", Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belrose JC, Noppens RR. Anesthesiology and cognitive impairment: a narrative review of current clinical literature. BMC Anesthesiol. 2019 Dec 27;19(1):241. doi: 10.1186/s12871-019-0903-7. PMID 31881996
- [Background] Daiello LA, Racine AM, Yun Gou R, Marcantonio ER, Xie Z, Kunze LJ, Vlassakov KV, Inouye SK, Jones RN, Alsop D, Travison T, Arnold S, Cooper Z, Dickerson B, Fong T, Metzger E, Pascual-Leone A, Schmitt EM, Shafi M, Cavallari M, Dai W, Dillon ST, McElhaney J, Guttmann C, Hshieh T, Kuchel G, Libermann T, Ngo L, Press D, Saczynski J, Vasunilashorn S, O'Connor M, Kimchi E, Strauss J, Wong B, Belkin M, Ayres D, Callery M, Pomposelli F, Wright J, Schermerhorn M, Abrantes T, Albuquerque A, Bertrand S, Brown A, Callahan A, D'Aquila M, Dowal S, Fox M, Gallagher J, Anna Gersten R, Hodara A, Helfand B, Inloes J, Kettell J, Kuczmarska A, Nee J, Nemeth E, Ochsner L, Palihnich K, Parisi K, Puelle M, Rastegar S, Vella M, Xu G, Bryan M, Guess J, Enghorn D, Gross A, Gou Y, Habtemariam D, Isaza I, Kosar C, Rockett C, Tommet D, Gruen T, Ross M, Tasker K, Gee J, Kolanowski A, Pisani M, de Rooij S, Rogers S, Studenski S, Stern Y, Whittemore A, Gottlieb G, Orav J, Sperling R; SAGES Study Group*. Postoperative Delirium and Postoperative Cognitive Dysfunction: Overlap and Divergence. Anesthesiology. 2019 Sep;131(3):477-491. doi: 10.1097/ALN.0000000000002729. PMID 31166241
- [Background] Lee SH, Lim SW. Risk factors for postoperative delirium after colorectal surgery: a systematic review and meta-analysis. Int J Colorectal Dis. 2020 Mar;35(3):433-444. doi: 10.1007/s00384-019-03498-6. Epub 2020 Jan 2. PMID 31897646
- [Background] Park SA, Tomimaru Y, Shibata A, Miyagawa S, Noguchi K, Dono K. Incidence and Risk Factors for Postoperative Delirium in Patients After Hepatectomy. World J Surg. 2017 Nov;41(11):2847-2853. doi: 10.1007/s00268-017-4079-3. PMID 28608014
- [Background] Saxena S, Maze M. Impact on the brain of the inflammatory response to surgery. Presse Med. 2018 Apr;47(4 Pt 2):e73-e81. doi: 10.1016/j.lpm.2018.03.011. Epub 2018 Apr 12. PMID 29656802
- [Background] Inoue R, Sumitani M, Ogata T, Chikuda H, Matsubara T, Kato S, Shimojo N, Uchida K, Yamada Y. Direct evidence of central nervous system axonal damage in patients with postoperative delirium: A preliminary study of pNF-H as a promising serum biomarker. Neurosci Lett. 2017 Jul 13;653:39-44. doi: 10.1016/j.neulet.2017.05.023. Epub 2017 May 11. PMID 28504118
- [Background] Alam A, Hana Z, Jin Z, Suen KC, Ma D. Surgery, neuroinflammation and cognitive impairment. EBioMedicine. 2018 Nov;37:547-556. doi: 10.1016/j.ebiom.2018.10.021. Epub 2018 Oct 19. PMID 30348620
- [Background] Evered LA, Chan MTV, Han R, Chu MHM, Cheng BP, Scott DA, Pryor KO, Sessler DI, Veselis R, Frampton C, Sumner M, Ayeni A, Myles PS, Campbell D, Leslie K, Short TG. Anaesthetic depth and delirium after major surgery: a randomised clinical trial. Br J Anaesth. 2021 Nov;127(5):704-712. doi: 10.1016/j.bja.2021.07.021. Epub 2021 Aug 28. PMID 34465469